CLINICAL TRIAL: NCT06987201
Title: Prospective, Crossover, Open Label Study to Evaluate the Effects of Vibration Anesthesia With DigiVibe on Pain in Subjects Undergoing Intramuscular Injections, Subcutaneous Injections, and Fingersticks (VIB-DIGI)
Brief Title: Effects of DigiVibe on Pain in Subjects Undergoing Intramuscular Injections, Subcutaneous Injections, and Fingersticks
Acronym: VIB-DIGI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: East Coast Institute for Research (Network)
Collaborators: Universal Axon Clinical Research, LLC (Unknown); Suthe Dermal (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: UACR-DIGI-01
Record Dates: First submitted 2025-05-09; First posted 2025-05-23 (Actual); Results first posted 2026-01-14 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2025-12

CONDITIONS: Healthy
Keywords: DigiVibe; Vibration Anesthesia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- No DigiVibe (No Intervention): Standard of Care
- DigiVibe (Experimental): DigiVibe Vibration Anesthesia
  Interventions: Device: DigiVibe Vibration Anesthesia

INTERVENTIONS:
Device: DigiVibe Vibration Anesthesia — DigiVibe Vibration Anesthesia
  Arms: DigiVibe

SUMMARY:
This is a single-center, unblinded, prospective, cross-over study. The study population will include twenty (n=20) healthy subjects (10 men and 10 women) over the age of 18 with a self-reported fear/dislike of needles. Subjects who qualify for the study based on the study inclusion and exclusion criteria and who consent to participate in the study will undergo two (2) intramuscular (IM) injections in the deltoid muscle, two (2) subcutaneous (SC) injections in the abdomen, and two (2) fingersticks with a lancing device in the middle finger. One injection in each location will be performed using with no intervention (as per standard of care) and the other injection in each location will be performed using the DigiVibe device.

DETAILED DESCRIPTION:
While the complete mechanisms of pain and pain diversion are not completely understood, DigiVibe locally targets the skin's pain receptors. Therefore, it is proposed that the vibrations from the DigiVibe device will counteract and/or lessen the pain around the injection site. This study will determine whether the use of DigiVibe during a procedure requiring injections provides greater reduction in pain than injections with no intervention (standard of care). This information will aid healthcare providers in selecting the best approach to management of pain in patients who must undergo injections that could cause pain and may benefit from additional pain reduction.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. BMI 18.5-29.9 kg/m2 (normal)
3. Self-reported fear/dislike of needles

Exclusion Criteria:

1. Chronic (daily) use of nonsteroidal anti-inflammatory drugs (NSAIDs) (i.e. ibuprofen, aspirin, naproxen, etc.), antiplatelet medications (i.e. clopidogrel, prasugrel, ticagrelor, cangrelor, cilostazol, etc), or anticoagulant medications (i.e. warfarin, dabigatran, rivaroxaban, apixaban, edoxaban, heparin, enoxaparin, fondaparinux, etc.)

   * Note: NSAIDs used as needed are not excluded as long as they are not used within 3 days of study screening and enrollment
2. Chronic (daily) use of analgesics (i.e. acetaminophen, NSAIDs [ie. ibuprofen, naproxen], opioids [ie. morphine, oxycodone, fentanyl], lidocaine, cannabinoids [ie. CBD, THC],)

   * Note: analgesics used as needed are not excluded as long as they are not used within 3 days of study screening and enrollment
3. Any condition in the opinion of the study investigator that would potentially confound the results of this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2025-08-04 (Actual); Primary Completion 2025-08-15 (Actual); Study Completion 2025-08-15 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Universal Axon Clinical Research, LLC, Doral, Florida, United States

IPD SHARING:
Plan to Share IPD: Yes
Only IPD used in the results publication
Supporting Information: Study Protocol, SAP, ICF
Time Frame: May 15, 2025 through July 31, 2025

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 1. Males and Females Age ≥ 18 years
  2. BMI 18.5-29.9 kg/m2 (normal)
  3. Self-reported fear/dislike of needles
Pre-assignment Details: 1. Males and Females Age ≥ 18 years
  2. BMI 18.5-29.9 kg/m2 (normal)
  3. Self-reported fear/dislike of needles
Groups:
- No DigiVibe (SOC), Then Digivibe: Participants received two rounds of injections with and without vibration anesthesia (DigiVibe) and completed Visual Analog Scale (VAS) pain scales immediately following the both rounds of injections. The first round of injections involved the Standard of Care (SOC) (injections without vibration anesthesia) with one subcutaneous abdomen (30G, 4mm needle with normal saline), one intramuscular deltoid (either 25G or 30G, 1 inch needles with normal saline), and one fingerstick (30G, 1.5 mm needle). After waiting 5 minutes, the DigVibe vibration anesthesia device was applied for 20 seconds (before and during lancing) and the second abdomen, deltoid, and fingerstick injections were administered.
Period: Overall Study
Arm/Group | No DigiVibe (SOC), Then Digivibe
Started | 20
SOC: Abdomen SC (30G, 4mm needle) | 20
DigiVibe: Abdomen SC (30G, 4mm needle) | 20
SOC: Deltoid IM (25G only, 1 inch needle) | 10
Digivibe: Deltoid IM (25G only, 1 inch needle) | 10
SOC: Deltoid IM (30G only, 1 inch needle) | 10
Digivibe: Deltoid IM (30G only, 1 inch needle) | 10
SOC: Fingerstick (30G, 1.5 mm needle) | 20
Digivibe: Fingerstick (30G, 1.5 mm needle) | 20
Completed | 20
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Cross-Over Trial of males and females ≥ 18 years old who have a normal BMI of 18.5-29.9 kg/m2, and a self-reported fear/dislike of needles.
Arm/Group | No DigiVibe (SOC), Then Digivibe
Number analyzed (Participants) | 20
Age, Continuous [Mean (Standard Deviation); unit: Years] — Age Population: Age of individuals who received injections without Digivibe and then with Digivibe
  Years | 37.5 (13.4)
Sex: Female, Male [Count of Participants; unit: Participants] — Sex Population: Sex of individuals who received injections without Digivibe and then with Digivibe
  Participants
    Female | 10
    Male | 10
Race (NIH/OMB) [Count of Participants; unit: Participants] — Race Population: Race of individuals who received injections without Digivibe and then with Digivibe
  Participants
    American Indian or Alaska Native | 0
    Asian | 0
    Native Hawaiian or Other Pacific Islander | 0
    Black or African American | 0
    White | 20
    More than one race | 0
    Unknown or Not Reported | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Ethnicity Population: Ethnicity of individuals who received injections without Digivibe and then with Digivibe
  Participants
    Hispanic or Latino | 19
    Not Hispanic or Latino | 1
    Unknown or Not Reported | 0
Height [Mean (Standard Deviation); unit: Inches] — Height Population: Height of individuals who received injections without Digivibe and then with Digivibe
  Inches | 308 (18.9)
Weight [Mean (Standard Deviation); unit: Lbs] — Weight of individuals who received injections without Digivibe and then with Digivibe
  Lbs | 157.5 (22.9)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m2] — BMI of individuals who received injections without Digivibe and then with Digivibe
  kg/m2 | 26 (2.4)
Systolic Blood Pressure (SBP) [Mean (Standard Deviation); unit: mmHg] — SBP of individuals who received injections without Digivibe and then with Digivibe
  mmHg | 115.4 (8.3)
Diastolic Blood Pressure (DBP) [Mean (Standard Deviation); unit: mmHg] — DBP of individuals who received injections without Digivibe and then with Digivibe
  mmHg | 71.1 (7.6)

OUTCOME MEASURES:

1. Primary Outcome: Mean Visual Analogue Scale (VAS) Pain Scale
Description: The original pain scores (Higher scores = worse pain) were represented by a grading scale of zero (0) to ten (10) on the VAS pain scale questionnaire. The mean in the values is represented by the mean of the original VAS scores without DigiVibe or with DigiVibe across all the participants and injection types.
Time Frame: 1 day
Population: Pain scores of individuals who acted as their own control after receiving 6 total injections and completed a Visual Analog Scale (VAS) pain scales immediately following the both rounds of injections (no DigiVibe compared to injections with DigiVibe).
Measure: Mean (95% Confidence Interval); unit: Units on a scale
Groups:
- No DigiVibe First (SOC), Then DigiVibe: Participants received two rounds of injections with and without vibration anesthesia (DigiVibe) and completed Visual Analog Scale (VAS) pain scales immediately following the both rounds of injections. The first round of injections involved the Standard of Care (SOC) (injections without vibration anesthesia) with one subcutaneous abdomen (30G, 4mm needle with normal saline), one intramuscular deltoid (either 25G or 30G, 1 inch needles with normal saline), and one fingerstick (30G, 1.5 mm needle). After waiting 5 minutes, the DigVibe vibration anesthesia device was applied for 20 seconds (before and during lancing) and the second abdomen, deltoid, and fingerstick injections were administered.
Arm/Group | No DigiVibe First (SOC), Then DigiVibe
Number analyzed (Participants) | 20
Units on a scale
  Mean VAS for Abdomen SC (30G, 4mm needle) - SOC | 3.75 [3.01 to 4.49]
  Mean VAS for Abdomen SC (30G, 4mm needle) - With DigiVibe | 1.10 [0.60 to 1.60]
  Mean VAS for total Deltoid (25G and 30G, 1 inch needle) - SOC | 3.85 [3.07 to 4.63]
  Mean VAS for total Deltoid (25G and 30G, 1 inch needle) - With DiVibe | 1.85 [1.24 to 2.46]
  Mean VAS for Deltoid (25G only, 1 inch needle) - SOC | 4.40 [3.22 to 5.58]
  Mean VAS for Deltoid (25G only, 1 inch needle) - With DigiVibe | 1.90 [0.76 to 3.04]
  Mean VAS for Deltoid (30G only, 1 inch needle) - SOC | 3.30 [2.18 to 4.42]
  Mean VAS for Deltoid (30G only, 1 inch needle) - With DigiVibe | 1.80 [1.06 to 2.54]
  Mean VAS for Fingerstick (30G, 1.5 mm needle) - SOC | 2.35 [1.72 to 2.98]
  Mean VAS for Fingerstick (30G, 1.5 mm needle) - With DigiVibe | 0.60 [0.13 to 1.07]
Statistical Analysis 1: Comparison: No DigiVibe First (SOC), Then DigiVibe; Test type: Other — Test for Difference Between Groups; p < 0.001, t-test, 2 sided; Mean Difference (Final Values) = -2.650, 95% CI 2-sided [-3.398 to -1.902]

ADVERSE EVENTS:
Time Frame: 1 day
Description: An adverse event (AE) is any untoward, undesired, or unplanned event in the form of signs, symptoms, disease, or laboratory or physiologic observations occurring in a person given a test article or in a clinical study.
Arm/Group | No DigiVibe (SOC), Then Digivibe
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 0/20

LIMITATIONS AND CAVEATS:
Lack of sham control and blinding.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-05-04): https://cdn.clinicaltrials.gov/large-docs/01/NCT06987201/Prot_SAP_000.pdf